CLINICAL TRIAL: NCT01746264
Title: Effect of Vitamin D Supplementation on Endothelial Function in Obese Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Seema Kumar, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-006349; UL1TR000135 (NIH)
Record Dates: First submitted 2012-11-16; First posted 2012-12-10 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Obesity; Endothelial Dysfunction; Vitamin D Deficiency
Keywords: Obesity; Endothelial dysfunction; Vitamin D deficiency
MeSH Terms: conditions — Obesity; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D3 (Experimental): Vitamin D3 supplementation at 100,000 IU once a month for 3 months
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D 3 at 100,000 IU once a month for 3 months
  Other Names: Cholecalciferol

SUMMARY:
Vitamin D deficiency has been linked to endothelial dysfunction in adults. Obese adolescents have a high prevalence of Vitamin D deficiency as well as evidence of endothelial dysfunction. Our hypothesis is that supplementation of Vitamin D deficient adolescents with Vitamin D would lead to improvement in endothelial dysfunction.

DETAILED DESCRIPTION:
Subjects had a brief screening visit with one of the study team members. Past medical history, current medications and a brief dietary history was taken. The dietary history was taken to assess calcium intake in a day and was obtained via the validated Short Calcium questionnaire. Blood pressure, heart rate as well as height,weight, waist and hip circumference measurement was obtained by study staff. In addition, a brief physical examination to determine Tanner stage was also completed. This involved examination of both breasts and genitalia for adolescent female and only genitalia in males. A physical activity questionnaire (IPAQ) was also administered by the study staff at this visit. A blood draw of 5 ml to measure plasma 25(OH) D, calcium, phosphorus was obtained as part of the screening visit. For girls who had started menstruating, a urine pregnancy test was also obtained.

After the screening visit eligible subjects had baseline biochemical tests and an endothelial function assessment. Study participants received a pill container with six total pills of vitamin cholecalciferol (D3) (1 pill = 50,000 IU), with directions to take two pills once a month (100,000 IU) at the same time for a period of 3 months. Compliance was assessed at the 3 month visit by counting the number of pills remaining in the container.

At 1 month, the subjects had tests for serum calcium and 25 hydroxy vitamin D levels. A urine test for random calcium to creatinine ratio was also obtained.

At 2 months, the serum calcium, 25 hydroxy vitamin D levels, and calcium to creatinine ratio tests were repeated.

At the end of 3 months, biochemical tests and an endothelial function assessment were repeated. Medical history, questionnaires, and the physical exam were also repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-18 years
2. BMI >95% for age and gender
3. 25 (OH) D levels less than 30 ng/ml

Exclusion Criteria:

1. 25 (OH) D levels >30 ng/mL
2. Serum calcium >10.4 mg/dL
3. Serum phosphorus > 4.7 mg/dl
4. Pregnancy or nursing
5. Current cancer
6. Patients on vitamin D3 supplementation exceeding 400 IU/day
7. Hypertension defined as Blood Pressure over the 95th percentile for age, gender and height
8. Dietary calcium intake exceeding 1500 mg/day
9. Hepatic or renal disorders
10. Type 1 or type 2 diabetes mellitus
11. Subjects receiving insulin, metformin, or oral hypoglycemic medications
12. Subjects with malabsorption disorders (celiac disease, cystic fibrosis, inflammatory bowel disease)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Kumar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Javed A, Kullo IJ, Balagopal PB, Kumar S. Effect of vitamin D3 treatment on endothelial function in obese adolescents. Pediatr Obes. 2016 Aug;11(4):279-84. doi: 10.1111/ijpo.12059. Epub 2015 Aug 14. PMID 26273791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between February 2013 and December 2013 at Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Vitamin D3
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilatation (FMD)
Description: Endothelial function was assessed by FMD, via a high-resolution Doppler ultrasonography examination of the right brachial artery. FMD was calculated as the maximal percentage increase in brachial artery diameter (BAD) from baseline after the release of cuff occlusion.
Time Frame: baseline, 3 months
Population: Data for one subject could not be included as the data on FMD was lost in the system and could not be retrieved.
Measure: Mean (Standard Deviation); unit: percentage increase in BAD
Arm/Group | Vitamin D3
Number analyzed (Participants) | 18
percentage increase in BAD
  Baseline FMD | 9.5 (3.52)
  3 months FMD | 10.4 (3.82)
Statistical Analysis 1: Comparison: Vitamin D3; P-value for change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.59, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: 25-hydroxy Vitamin D (25[OH]D) Levels
Description: 25(OH)D was measured using liquid chromatography-tandem mass spectrometry. Total 25(OH)D concentrations of each sample was calculated using internal standard, 25(OH)D_2 and 25(OH)D_3.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
nmol/L
  baseline 25(OH)D | 55.9 (12.2)
  3 months 25(OH)D | 86.9 (16.7)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow up visit; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Cholesterol
Description: Total cholesterol levels were measured by an enzymatic colorimetric assay.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
mmol/L
  baseline | 3.69 (0.71)
  3 months | 4.03 (0.87)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Triglycerides
Description: Total triglyceride levels were measured by an enzymatic colorimetric assay.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
mmol/L
  Baseline | 1.19 (0.57)
  3 months | 1.58 (0.81)

5. Secondary Outcome: Body Mass Index
Description: Body Mass Index (BMI) is a health index for comparing weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared. The body mass index is an indication if a person is at a suitable weight for his height on an approximation of body fat. A body mass index of under 20 is considered to be underweight, while a body mass index between 20 to 25 is considered healthy. A body mass index in the range of 25 to 30 is regarded as overweight. A body mass index over 30 is regarded as obese.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
kg/m^2
  baseline | 36.1 (6.03)
  3 months | 36.4 (6.11)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: International Physical Activity Questionnaire (IPAQ) Short Form Score
Description: The IPAQ short form used asked 7 questions about activities in the last 7 days, covering vigorous physical activities, moderate activities, walking, and sitting, asking for days per week, hours per day or minutes per day. The score is reported in metabolic equivalent (MET)-minutes per week. Possible scores could range from 0 (inactive) to greater than 3000 MET-minutes/week (highly active). The definition of high activity was vigorous intensity activity on at least 3 days achieving a minimum total activity of at least 1500 MET-minutes/week OR 7 days of any combination of walking, moderate-intensity or vigorous-intensity activities achieving a minimum total physical activity of at least 3000 MET-minutes/week. Therefore a score of > 3000 MET-minutes/week was possible.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: MET-minutes per week
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
MET-minutes per week
  baseline | 1786.6 (1506.2)
  3 months | 2799.1 (3834.6)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3-month follow-up; Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Calcium Intake Per Day
Description: Calcium intake was measured using the validated Short Calcium Questionnaire (SCQ). This questionnaire is in the form of an spreadsheet, and asks the participant to enter the number of servings per week of various food items and vitamin or mineral supplements. The spreadsheet calculates the daily calcium intake (mg/day) from the data entered.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
mg/day
  baseline | 1102.7 (304.3)
  3 months | 975.5 (282.2)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Serum Parathyroid Hormone (PTH)
Description: A parathyroid hormone (PTH) blood test measures the level of parathyroid hormone in the blood. This test is used to help identify hyperparathyroidism, to find the cause of abnormal calcium levels, or to check the status of chronic kidney disease. PTH controls calcium and phosphorus levels in the blood. PTH was measured by a two-site chemiluminescent immunometric assay.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
pmol/L
  baseline | 4.1 (1.6)
  3 months | 3.3 (1.1)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.0123, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Fasting Glucose
Description: Plasma glucose was measured by hexokinase enzymatic assay.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
mmol/L
  baseline | 4.9 (0.28)
  3 months | 4.97 (0.26)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Fasting Insulin
Description: Serum insulin was measured using commercial electrochemiluminescence immunoassay kits.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
pmol/L
  baseline | 225.71 (127.93)
  3 months | 245.16 (150.01)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.27, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Homeostatic Model Assessment of Insulin Resistance Index (HOMA-IR)
Description: This calculation measures insulin resistance, and requires U.S. standard units. The healthy range is 0.5 to 1.4. Less than 1.0 means the subject is insulin-sensitive, which is optimal. Above 1.9 indicates early insulin resistance. Above 2.9 indicates significant insulin resistance. The HOMA-IR was calculated as: HOMA-IR = fasting serum glucose (mmol/L) x fasting insulin (mU/mL)/22.5.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: index of beta cell function
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
index of beta cell function
  baseline | 7.11 (4.18)
  3 months | 7.9 (5.1)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: High Sensitivity C-reactive Protein (Hs-CRP)
Description: A high-sensitivity C-reactive protein (hs-CRP) test may be used to help evaluate an individual for risk of cardiovascular disease (CVD). C-reactive protein (CRP) is a protein that increases in the blood with inflammation. Studies have suggested that a persistent low level of inflammation plays a major role in atherosclerosis, the narrowing of blood vessels due to build-up of cholesterol and other lipids, which is often associated with CVD. The hs-CRP test accurately measures low levels of C-reactive protein to identify low but persistent levels of inflammation and thus helps predict a person's risk of developing CVD. hs-CRP was measured using particle-enhanced immunonephelometry.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
nmol/L
  baseline | 47.62 (35.43)
  3 months | 40 (25.7)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.33, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Low-density Lipoprotein Cholesterol (LDL) Cholesterol Levels
Description: The test for low-density lipoprotein cholesterol is used as part of a lipid profile to predict an individual's risk of developing heart disease. A desirable level is <3.36 mmol/L; borderline high is 3.36 - 4.11 mmol/L; high is >/= 4.14 mmol/L. LDL cholesterol was calculated as: LDL = Total cholesterol - HDL cholesterol - Triglycerides/5.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
mmol/L
  baseline | 1.95 (0.66)
  3 months | 2.15 (0.81)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: High Density Lipoprotein (HDL) Cholesterol Levels
Description: Total HDL cholesterol levels were measured by an enzymatic colorimetric assay. The test for high-density lipoprotein cholesterol (HDL-C) is used along with other lipid tests to screen for unhealthy levels of lipids and to determine the risk of developing heart disease. If a subject has a negative risk factor, a desirable HDL level would be >/= 1.55 mmol/L.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
mmol/L
  baseline | 1.2 (0.28)
  3 months | 1.16 (0.23)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Urine Calcium to Creatinine Ratio
Description: Urine calcium/creatinine ratio (unit mg/g) on random urine sample was calculated by dividing calcium in mg by creatinine in g.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Vitamin D3
Number analyzed (Participants) | 19
mg/g
  baseline | 67.8 (59.2)
  3 months | 87.7 (73.2)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.32, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Reactive Hyperemia Index (RHI)
Description: The cuff of a sphygmomanometer was placed on the forearm and inflated to 50 mm Hg above the participant's systolic blood pressure for a period of 5 min. The increase in resting brachial blood flow was calculated as the maximum flow recorded in the first 15 seconds after cuff deflation and expressed as a percentage increase from baseline reactive. Higher values are considered normal or improved endothelial function.
Time Frame: baseline, 3 months
Population: Data for one subject could not be included as the data on RHI was lost in the system and could not be retrieved.
Measure: Mean (Standard Deviation); unit: percentage increase in blood flow
Arm/Group | Vitamin D3
Number analyzed (Participants) | 18
percentage increase in blood flow
  baseline | 449.3 (243.5)
  3 months | 513.9 (325.6)
Statistical Analysis 1: Comparison: Vitamin D3; Change from baseline to 3 month follow-up; Test type: Superiority or Other; p = 0.47, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Vitamin D3
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes